CLINICAL TRIAL: NCT00515684
Title: Corneal Thinning During Topical Bevacizumab Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Side effect can increase the risk of the research
Sponsor: Yonsei University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 4-2006-0234
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Corneal Neovascularization
MeSH Terms: conditions — Corneal Neovascularization | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bevacizumab (Avastin)

SUMMARY:
The purpose of this study is to determine whether topical bevacizumab is safe or not when used in corneal neovascularization for long term period.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of corneal neovascularization
* must be able to apply eyedrop

Exclusion Criteria:

* have active keratitis

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Woo Kim, M.D., Principal Investigator — Severance hospital, Seoul , Korea
Locations (1):
- Severance hospital, Seoul, South Korea